CLINICAL TRIAL: NCT03453099
Title: Modifiable Factors Affecting the Dose of Propofol Required for Anaesthetic Induction
Brief Title: MAPD: Modifiable Factors Affecting Propofol Dosing
Status: Completed | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 00001
Record Dates: First submitted 2018-02-13; First posted 2018-03-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia
Keywords: propofol; anaesthetic dose; sleep; caffeine; anxiety; induction
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Any ASA I or II patients scheduled for elective day case general anaesthesia at Chelsea & Westminster Hospital, involving a standard propofol-fentanyl induction regimen, aged between 18-65 years . See specific exclusion criteria below.
  Interventions: Other: Preoperative Questionnaires; Other: Postoperative Subjective Pain Scores

INTERVENTIONS:
Other: Preoperative Questionnaires — The participants will be asked to complete 5 questionnaires:
  1. An abbreviated version of the Caffeine Assessment Tool (CAT)
  2. Sleep Questionnaire (SQ)
  3. Surgical Fear Questionnaire (SFQ)
  4. WHO Alcohol AUDIT Tool
  5. WHO Smoking Questionnaire
  They will also be asked to complete a demographics sheet
  All participants will undergo standard anaesthetic induction, a research participant will observe the dose of propofol and time taken for loss of consciousness
Other: Postoperative Subjective Pain Scores — After the operation, participants will be provide with a scale from 1-10 in which to rate their pain at rest and whilst coughing. This will be undertaken at 1hr postoperatively.

SUMMARY:
The investigators aim to understand the effect of a caffeine intake, sleep habits, anxiety about surgery, alcohol intake and smoking status upon the dose of the anaesthetic drug, propofol, required for anaesthetic induction.

DETAILED DESCRIPTION:
The investigators hypothesise that modifiable environmental factors may cause reversible changes in a patients neurobiology which affect their responsiveness to anaesthetic drugs. Such factors may include chronic caffeine intake, chronic sleep deprivation, acute anxiety about surgery, alcohol intake and smoking. Investigation of the relationship between such factors and the dose of anaesthetic required for loss of consciousness may not only allow for better prediction of dose requirements but may also allow for optimisation of patients prior to undergoing general anaesthesia with a view to decreasing anaesthetic dose requirements and the complications associated with this.

To address this questions, the investigators will be asking patients admitted for any day case surgery at Chelsea & Westminster hospital to complete five short questionnaires and a demographic sheet addressing 1) Caffeine intake 2) Sleep habits 3) Anxiety about the operation 4) Alcohol intake 5) Smoking status.

This will then be compared to the amount of the anaesthetic drug Propofol required and the time taken to induce loss of consciousness prior to surgery. Loss of consciousness will be measured subjectively by loss of eye opening response and loss of verbal response when a patient is asked to count upwards from 1.

The investigators also wish to investigate whether these same 5 factors affect patient reported postoperative pain and analgesia requirements. As such the investigators will also ask participants to rate their level of pain whilst at rest and whilst coughing at 1 hour after the operation. We will also record how much analgesia is requested and received in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

ASA I or II patients scheduled for elective day case general anaesthesia with Laryngeal Mask Airway (LMA) airway insertion and a standard propofol-fentanyl induction, aged between 18-65 years at Chelsea & Westminster Hospital.

Exclusion Criteria

1. Pregnancy
2. Neurological disease
3. Substance abuse
4. Cardiac disease
5. Renal disease
6. Obesity

Additional exclusion criteria include:

1. Any patient requiring adjunctive analgesia including local/epidural/spinal anaesthesia.
2. Any patient requiring an anesthetic induction regime other than propofol-fentanyl (inc. administration of benzodiazepines or other strong opioids).
3. Any patient who does not receive a standard anaesthetic induction regime due to clinical need

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient scheduled for day case general anasethesia at Chelsea & Westminster hospital who satisfy the listed inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
The dose of propofol required for anaesthetic induction | 10 minutes
  Propofol will be administered at a rate of 20mg every 10 seconds by the Anaesthetist (as per national guidelines) and a member of the research team will passively record the dose of drug and the time taken for loss of consciousness as defined by a lack of eye opening and a lack of verbal response

SECONDARY OUTCOMES:
Postoperative patient reported pain scores | 5 minutes
  Participants will rate their level of postoperative pain whilst at rest and whilst coughing 1hr postoperatively using a Visual Analogue Scale (1-10)

OTHER OUTCOMES:
Postoperative Analgesia Requirements | 5 minutes
  A member of the research team will passively record the amount of analgesia required at 1hr postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No